CLINICAL TRIAL: NCT04081584
Title: Trans-abdominal Fetal Pulse Oximetry: Tissue Light Scattering
Status: Terminated | Type: Observational
Why Stopped: COVID-19
Sponsor: Raydiant Oximetry, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ISS
Record Dates: First submitted 2019-09-03; First posted 2019-09-09 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Fetal Distress
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: ISS Device — The ISS Device (commercial and prototype) is used to measure tissue light scattering.

SUMMARY:
This study is being conducted to study light scattering properties of maternal-fetal tissue.

DETAILED DESCRIPTION:
The ISS customized commercial frequency domain oximeter is used to obtain light scattering information from the maternal abdomen for 10-20 minutes preoperatively and postoperatively in subjects who are having a scheduled C-section.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women with singleton pregnancies, vertex or breech presentation, scheduled for non-emergent cesarean delivery, including cesarean delivery for failure to progress with reassuring electronic fetal heart rate tracing
2. Age greater than or equal to 18 years of age.
3. Healthy women at equal to or greater than 36 weeks gestation undergoing non-emergency cesarean delivery
4. Spinal or epidural anesthesia

Exclusion Criteria:

1. Emergency cesarian delivery
2. Non-reassuring fetal heart rate tracing
3. Less than 18 years of age
4. Multiple gestation (twins, triplets)
5. Presentation other than vertex or breech
6. Less than 36 weeks of gestation
7. General anesthesia

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing a C-Section
Study Population: Women with singleton pregnancies of 36 weeks gestation or more undergoing c-section.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Optical signal from maternal and fetal tissues | Peri-operative
  The study of light scattering through maternal/fetal tissue and through maternal tissue alone and newborn tissue alone using a commercial frequency domain oximeter and 2nd generation prototype.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No